CLINICAL TRIAL: NCT02305082
Title: Fast-track Giant Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, PHD student, Bispebjerg Hospital
Other Study IDs: Fast-track-hernia-bbh
Record Dates: First submitted 2014-11-11; First posted 2014-12-02 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fast-track group: Patients treated according to the enhanced recovery pathway. This group is examined prospectively.
  Interventions: Other: Fast-track group
- Control group: Patients treated according to the historic recovery pathway. This group is examined retrospectively.

INTERVENTIONS:
Other: Fast-track group — Enhanced recovery after surgery pathway. Postoperatively, a set of well-defined discharge criteria will be assessed daily at 9:00 and 15:00, as well as pain, nausea, time to flatus, saturation and drain production.
  Groups: Fast-track group

SUMMARY:
The implementation of an enhanced recovery pathway after giant ventral hernia repair, including preoperative high-dose steroid is examined prospectively and compared with a group of historic controls.

DETAILED DESCRIPTION:
All patients operated on for a large incisional hernia are treated according to the study protocol. Patients are given high-dose glucocorticoid preoperative and the aim is to discharge patients at postoperative day 3.

Morbidity, length of stay, pain, nausea and pulmonary function are among registered outcomes compared with a historic control group.

ELIGIBILITY:
Inclusion Criteria:

* Horizontal fascia defect > 10 cm on computed tomography scan
* Planned elective open incisional hernia repair

Exclusion Criteria:

* Known allergy against glucocorticoid treatment
* Insulin-treated diabetes
* Gastric ulcer diagnosed within four weeks preoperative
* Steroid-treated immune disease
* Planned intestinal anastomosis concomitant to hernia repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled to undergo elective incisional hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Time to discharge | Participants will be followed for the duration of hospital stay, an expected average of 72 hours
  Time from surgery to discharge [Hours].

SECONDARY OUTCOMES:
Fatigue | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Preoperative and twice daily (9 and 15) postoperative. Measured by a numerical rating scale (1 = No fatigue, 5 = Exhausted).
Pain from supine to standing | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Preoperative and twice daily (9 and 15) postoperative. Measured by a numerical rating scale (1 = No pain, 5 = Intolerable pain)
Pain when walking 6 meters | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Preoperative and twice daily (9 and 15) postoperative. Measured by a numerical rating scale (1 = No pain, 5 = Intolerable pain)
Nausea | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Preoperative and twice daily (9 and 15) postoperative. Measured by a numerical rating scale (1 = No nausea, 5 = Intolerable nausea)
Time to bowel function | For the duration of postoperative hospital stay, an expected average of 72 hours
  The time to bowel function [hours] will be registered for each participant
Vomiting episodes | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  The daily number of vomiting episodes will be registered for each participant
Continuous transcutaneous saturation | From surgery to postoperative day 3 at 12 pm
  Continuous transcutaneous oxygen saturation (percentage), measured by Pulsox 300i (C) (Konica Minolta, Osaka, Japan)
C-reactive protein from venous blood sample | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Daily C-reactive protein measured in a venous blood sample.
Ear temperature | Preoperative and for the duration of hospital stay, an expected average of 3 days
  Ear temperature (celsius degree) measured daily at 9 and 15.
Detailed reason for not being discharged if criteria are otherwise fulfilled | From surgery and for the duration of hospital stay, an expected average of 3 days
  The reason(s) for participants not being discharged if discharge criteria are otherwise fulfilled.
Daily wound drain production | From surgery and for the duration of hospital stay, an expected average of 3 days
  Daily registration of the fluid volume [milliliters] in the wound drains postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Jensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark